CLINICAL TRIAL: NCT03849118
Title: A Confirmatory, Prospective, Open-label, Multi-centre Phase 3 Study to Evaluate Diagnostic Performance of Zirconium-labelled Girentuximab to Non-invasively Detect ccRCC by PET/CT Imaging in Patients With Indeterminate Renal Masses
Brief Title: 89Zr-TLX250 for PET/CT Imaging of ccRCC- ZIRCON Study
Acronym: 89ZR-TLX250
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Telix Pharmaceuticals (Innovations) Pty Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 89Zr-TLX250-003
Record Dates: First submitted 2019-01-29; First posted 2019-02-21 (Actual); Results first posted 2024-05-17 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Clear Cell Renal Cell Carcinoma
Keywords: clear cell renal cell carcinoma; PET/CT imaging; 89Zr-girentuximab
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Intervention Model Description: diagnostic, confirmatory, prospective, multi-centre
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 89Zr-girentuximab (Experimental): A single administration of 37 Megabecquerel (MBq) (±10%) 89Zr-girentuximab, containing a mass dose of 10 mg of girentuximab, followed by a diagnostic scan on Day 5 ± 2 days after administration.
  Interventions: Diagnostic Test: 89Zr-girentuximab

INTERVENTIONS:
Diagnostic Test: 89Zr-girentuximab — Single IV administration on Day 0, followed by diagnostic scan on Day 5 +/- 2 days.
  Other Names: 89Zr-TLX250; 89Zr-DFO-TFP-girentuximab (GTX)

SUMMARY:
89Zr-TLX250 is under clinical development as a diagnostic agent targeting clear cell renal cell carcinoma.

DETAILED DESCRIPTION:
This is a confirmatory, prospective, open-label, multi-centre phase 3 study to evaluate sensitivity and specificity of 89Zr-TLX250 Positron Emission Tomography/Computed Tomography (PET/CT) imaging to non-invasively detect clear cell renal cell cancer (ccRCC) in adult patients with indeterminate renal masses (IRM), scheduled for partial or total nephrectomy.

Patients, will be recruited in 12-15 renal cancer care specialist centres, who have access to state-of-the-art PET/CT imaging equipment.

The study involves a single administration of 89Zr-TLX250. Imaging will then be conducted 5 +/-2 days post administration. The partial/total nephrectomy will then be performed at institutional discretion any time following the PET/CT imaging visit, but no later than 90 days post administration of 89Zr-TLX250. Histological tumour samples will be prepared and used for histological diagnosis of the renal mass (ccRCC or non-ccRCC) read by a central laboratory.

On Day 5 +/-2 post study drug administration, an abdominal PET/CT imaging will be obtained. In patients, in which unexpected evidence for disseminated disease is observed, PET/CT imaging may be extended to complete whole body imaging(vertex of skull to toe) at the discretion of the investigator.

Image data analyses will be performed by a central image core lab. Qualitative visual analysis (presence or absence of localised 89Zr-TLX250 uptake inside or in vicinity of renal lesion, as seen on contrast-enhanced CT or MRI), will be used to assess test performance or 89Zr-TLX-250 PET/CT imaging to non-invasively detect ccRCC, using histological results from the central histological reference laboratory as standard of truth.

ELIGIBILITY:
Inclusion Criteria:

1. Written and voluntarily given Informed Consent
2. Male or female ≥18 years of age
3. Imaging evidence of a single indeterminate renal mass of ≤7cm in largest diameter (tumour stage cT1) , on CT or MRI with and without contrast agent, suspicious for ccRCC
4. Scheduled for lesion resection as part of regular diagnostic work-up within 90 days from planned 89Zr-TLX250 administration
5. Negative serum pregnancy tests in female patients of childbearing potential (at Screening and within 24 hours prior to receiving investigational product)
6. for patients included in France only, verification and confirmation of their affiliation with a social security
7. Sufficient life expectancy to justify nephrectomy
8. Consent to practice double-barrier contraception until a minimum of 42 days after 89Zr-TLX250 administration

Exclusion Criteria:

1. Bioptic procedure (rather than a partial or total nephrectomy) planned for histological species delineation of IRM
2. Renal mass known to be a metastasis of another primary tumour
3. Active non-renal malignancy requiring therapy during the time frame of the study participation
4. Chemotherapy, radiotherapy or immunotherapy within 4 weeks prior to the planned administration of 89Zr-TLX250 or continuing adverse effects (> grade 1) from such therapy (Common Terminology Criteria for Adverse Events (CTCAE, Version 5.0)
5. Planned antineoplastic therapies (for the period between administration of 89 Zr-TLX250 and imaging)
6. Exposure to murine or chimeric antibodies within the last 5 years
7. Previous administration of any radionuclide within 10 half-lives of the same
8. Serious non-malignant disease (e.g. psychiatric, infectious, autoimmune or metabolic) that may interfere with the objectives of the study or within the safety of compliance of the subjects as judged by the Investigator
9. Mental impairment that may compromise the ability to give Informed Consent and comply with the requirements of the study
10. Exposure to any experimental diagnostic or therapeutic drug within 30 days from the date of planned administration of 89Zr-TLX250
11. Women who are pregnant or breastfeeding
12. Known hypersensitivity to Girentuximab or DFO (Desferrioxamine)
13. Renal insufficiency with glomerular filtration rate (GFR) ≤ 60 millilitres/min/1.73m2
14. Vulnerable patients (e.g being in detention)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2019-08-15 (Actual); Primary Completion 2022-10-20 (Actual); Study Completion 2022-11-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard Gurney, MD, Principal Investigator — Macquarie University Hospital; Francoise Brodere, MD, Principal Investigator — University Hospital ICO, Nantes, France; Peter Mulders, MD, Principal Investigator — Radboud University Medical Center; Marcel Stokkel, MD, Principal Investigator — The Netherlands Cancer Institute; Declan Murphy, MD, Principal Investigator — Victorian Comprehensive Cancer Centre; Andrew Scott, MD, Principal Investigator — Olivia Newton John Cancer Research Center, Austin Hospital; Simon Wood, MD, Principal Investigator — Princess Alexander Hospital; Mark Frydenberg, MD, Principal Investigator — Cabrini Hospital; David Chan, Principal Investigator — Royal North Shore Hospital; Jean-Christophe Bernhard, MD, Principal Investigator — CHU de Bordeaux, Groupe Hospitalier Pellegrin; Pierre Olivier, MD, Principal Investigator — CHRU de Nancy - Hôpitaux de Brabois; Linda Heijmen, MD, Principal Investigator — Leiden University Medical Centre; Martin Geert Steffens, MD, Principal Investigator — Isala; Karolien Goffin, MD, Principal Investigator — Universitair Ziekenhuis Leuven; Carlos Artigas Guix, MD, Principal Investigator — Instutit Jules Bordet; Nicolas Lumen, MD, Principal Investigator — University Ghent; Sumer Baltaci, MD, Principal Investigator — Ankara University; Bulent Akdogan, MD, Principal Investigator — Ankara Hacettepe University; Bulent Onal, MD, Principal Investigator — Istanbul University - Cerrahpasa; Tamer Aksoy, MD, Principal Investigator — Istanbul Training and Research Hospital
Locations (31):
- United States (9):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - University of California, Los Angeles Campus,, Los Angeles, California
  - Emory University, Atlanta, Georgia
  - Johns Hopkins University Hospital, Baltimore, Maryland
  - Advanced Molecular Imaging & Therapy, LLC, Glen Burnie, Maryland
  - Barbara Ann Karmanos Cancer Hospital, Detroit, Michigan
  - Washington University St Louis, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - SEATTLE CANCER CARE ALLIANCE, University of Washington, Seattle, Washington
- Australia (7):
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Macquarie University Hospital, Sydney, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Austin Health, Heidelberg, Victoria
  - Victorian Comprehensive Cancer Centre, Melbourne, Victoria
  - Cabrini Hospital, Melbourne, Victoria
- Belgium (2):
  - Institute Jules Bordet, Brussels
  - University Hospital Leuven (UZ Leuven), Leuven
- Canada (3):
  - Centre De Recherche Centre hospitalier de l/Universite de Montreal (CrCHUM ), Montreal, Quebec
  - Jewish General Hopsital, Montreal, Quebec
  - CHU de Québec - Université Laval - L'Hôtel-Dieu de Québec, Québec
- France (3):
  - CHU de Bordeaux, Groupe hospitalier Pellegrin, Bordeaux
  - CHRU de Nancy, Hopitaux de Brabois, Nancy
  - Nantes University Hospital Hotel-Dieu, Nantes
- Netherlands (2):
  - Netherlands Cancer Institute, Amsterdam
  - Radboud University Medical Centre, Nijmegen
- Turkey (Türkiye) (4):
  - Ankara University Medical Faculty Hospital, Ankara
  - Hacettepe University Faculty of Medicine, Ankara
  - Istanbul Training and Research Hospital, Istanbul
  - Istanbul University Cerrahpasa Medical Faculty, Istanbul
- Royal Free London NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chowdhury A, Morgat C, Bailly C, Sunderland J, Graves SA, Scott AM, Baker S, Holman BF. Radiation protection considerations with [89Zr]Zr-girentuximab PET and surgery. EJNMMI Res. 2025 May 23;15(1):59. doi: 10.1186/s13550-025-01247-1. PMID 40408016
- [Derived] Shuch B, Pantuck AJ, Bernhard JC, Morris MA, Master V, Scott AM, van Praet C, Bailly C, Onal B, Aksoy T, Merkx R, Schuster DM, Lee ST, Pandit-Taskar N, Fan AC, Allman P, Schmidt K, Tauchmanova L, Wheatcroft M, Behrenbruch C, Hayward CRW, Mulders P. [89Zr]Zr-girentuximab for PET-CT imaging of clear-cell renal cell carcinoma: a prospective, open-label, multicentre, phase 3 trial. Lancet Oncol. 2024 Oct;25(10):1277-1287. doi: 10.1016/S1470-2045(24)00402-9. Epub 2024 Sep 10. PMID 39270701

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 89Zr-girentuximab
Started | 300
Completed | 275
Not Completed | 25

BASELINE CHARACTERISTICS:
Groups:
- 89Zr-girentuximab: A single administration of 37 MBq (±10%) 89Zr-TLX250, containing a mass dose of 10 mg of girentuximab followed by a diagnostic scan on Day 5 ± 2 days
Arm/Group | 89Zr-girentuximab
Number analyzed (Participants) | 300
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 176
  >=65 years | 124
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86
  Male | 214
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaskan Native | 0
  Asian | 9
  Black or African American | 13
  Native Hawaiian or Other Pacific Islander | 0
  White | 277
  Missing | 1
Region of Enrollment [Number; unit: participants]
  Canada | 6
  Netherlands | 38
  Turkey | 29
  Belgium | 29
  United States | 113
  United Kingdom | 1
  Australia | 35
  France | 45
  Spain | 4

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity and Specificity of Qualitative Assessment of PET/CT Imaging With 89Zr-TLX250 to Noninvasively Detect ccRCC in Patients With Indeterminate Renal Masses, Using Histology as Standard of Truth.
Description: This outcome was evaluated on all patients by using a PET/CT machine to determine the uptake of the Zr89 radiotracer within the renal lesion. This was compared against the histological determination of the lesion type following resection of the lesion
Time Frame: Diagnostic PET/CT scan on Day 5 ± 2 days post 89Zr-TLX250 administration. Histological confirmation of the material from nephrectomy conducted within 90 days post 89Zr-TLX250 administration served as standard of truth.
Population: The overall number of participants analyzed consisted of all enrolled patients who had evaluable PET/CT imaging and a confirmed histopathology diagnosis. This number (284) is lower than the baseline participants (of 300) as 16 patients did not have both of these data points.
Measure: Count of Participants; unit: Participants
Groups:
- 89Zr-girentuximab: Single diagnostic administration, followed by a diagnostic scan on Day 5 ± 2 days.
Arm/Group | 89Zr-girentuximab
Number analyzed (Participants) | 284
Participants
  True negative | 84
  False positive | 11
  False negative | 30
  True Positive | 159

ADVERSE EVENTS:
Time Frame: 3 years
Groups:
- Adverse Events Information: The safety analysis set (SAF) consisted of all patients who received 89Zr-TLX250.
Arm/Group | Adverse Events Information
All-Cause Mortality (participants affected / at risk) | 2/300
Serious Adverse Events (participants affected / at risk) | 26/300
Other Adverse Events (participants affected / at risk) | 86/300
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adverse Events Information (N=300)
Anemia (Blood and lymphatic system disorders) | 1
Tachycardia (Cardiac disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 1
Hemoperitoneum (Gastrointestinal disorders) | 1
Intestinal Obstruction (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Retroperitoneal Effusion (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1
Death (General disorders) | 1
Multiple organ dysfunctional syndrome (General disorders) | 1
Ischemic Hepatitis (Hepatobiliary disorders) | 1
Hematoma Infection (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Klebsiella Infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Arterial Injury (Injury, poisoning and procedural complications) | 1
Post procedural bile leak (Injury, poisoning and procedural complications) | 1
Post procedural complication (Injury, poisoning and procedural complications) | 1
Post procedural hematuria (Injury, poisoning and procedural complications) | 1
Post procedural hemorrhage (Injury, poisoning and procedural complications) | 7
Post procedural hypotension (Injury, poisoning and procedural complications) | 1
Procedural pain (Injury, poisoning and procedural complications) | 1
Procedural pneumothorax (Injury, poisoning and procedural complications) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Hypovolemia (Metabolism and nutrition disorders) | 1
Hematoma muscle (Musculoskeletal and connective tissue disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 2
Acute kidney injury (Renal and urinary disorders) | 1
Renal Impairment (Renal and urinary disorders) | 1
Subcapsular renal hematoma (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 2
Urinoma (Renal and urinary disorders) | 1
Acute pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 1
Arteriosclerosis (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Adverse Events Information (N=300)
Abdominal Pain (Gastrointestinal disorders) | 5
Constipation (Gastrointestinal disorders) | 8
Diarrhea (Gastrointestinal disorders) | 8
Nausea (Gastrointestinal disorders) | 11
Vomiting (Gastrointestinal disorders) | 6
Procedural pain (Injury, poisoning and procedural complications) | 11
Hypertension (Vascular disorders) | 6
Headache (Nervous system disorders) | 9
Fatigue (General disorders) | 8
Pain (General disorders) | 7
Urinary tract infection (Infections and infestations) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If the Study is a Multi-center Study, then the Institution agrees that no publication of the study results may be made until publication of the results of the multi-center study or 2 years after study completion, whichever is the sooner.

DOCUMENTS (2):
  • Study Protocol (2022-04-01): https://cdn.clinicaltrials.gov/large-docs/18/NCT03849118/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-13): https://cdn.clinicaltrials.gov/large-docs/18/NCT03849118/SAP_001.pdf